CLINICAL TRIAL: NCT05440123
Title: Bronchopulmonary Cancer Screening Program and Primary Cardiovascular Prevention, Early Management of COPD and Smoking Cessation
Brief Title: Experimentation With Screening for Bronchopulmonary Cancer and Primary Cardiovascular Prevention, Early Management of COPD and an Offer Exempted From Smoking Cessation
Acronym: LUMASCAN-2
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: LUMASCAN-2
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: the Rate of Participation in Screening for PBC
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- bronchopulmonary cancer: The screening program includes performing a low-dose chest CT scan (STBD), spirometry, blood sampling (biobank + screening for cardiovascular risk factors) on inclusion, at 1 year and at 2 years. Subsequently, a telephone interview will be scheduled for 3 years to collect medical information, for a total follow-up period of 5 years. At each visit, a structured offer of smoking cessation will be proposed and a collection of the quality of life will be carried out. Each year, a telephone call from participants will be scheduled in order to maximize participation.
  For subjects presenting with anomalies suggestive of PBC on the STBD, a consultation in pneumo-oncology will be planned with management corresponding to routine care.
  Interventions: Other: screening for bronchopulmonary cancer

INTERVENTIONS:
Other: screening for bronchopulmonary cancer — The screening program includes performing a low-dose chest CT scan (STBD), spirometry, blood sampling (biobank + screening for cardiovascular risk factors) on inclusion, at 1 year and at 2 years. Subsequently, a telephone interview will be scheduled for 3 years to collect medical information, for a total follow-up period of 5 years. At each visit, a structured offer of smoking cessation will be proposed and a collection of the quality of life will be carried out. Each year, a telephone call from participants will be scheduled in order to maximize participation

SUMMARY:
The study consists of recruiting a target population by sending a letter from the Regional Center for Cancer Screening in Ile de France.

In the screening program, a battery of examinations will be carried out at inclusion, one year, 2 years, 3 years, 4 years and 5 years.

DETAILED DESCRIPTION:
The patients will be recruited by correspondence by by sending a letter from the Regional Center for Cancer Screening in Ile de France.

When the patient has agreed to participate, a screening program will be carried out The screening program includes performing a low-dose chest CT scan (STBD), spirometry, blood sampling (biobank + screening for cardiovascular risk factors) on inclusion, at 1 year and at 2 years. Subsequently, a telephone interview will be scheduled for 3 years to collect medical information, for a total follow-up period of 5 years. At each visit, a structured offer of smoking cessation will be proposed and a collection of the quality of life will be carried out. Each year, a telephone call from participants will be scheduled in order to maximize participation

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* Age: 55 to 74 years old
* Smokers at more than 20 pack-years weaned for less than 15 years
* Affiliated to a social security organization

Exclusion Criteria:

* Presence of signs of PBC
* Subjects with a personal history of PBC of less than 5 years or under treatment
* Presence of serious comorbidities involving the vital prognosis at 6 months
* Subjects who have already benefited from a chest CT scan less than one year old.
* Refusal to participate in the study
* Absence of exposure to tobacco or insufficient exposure to tobacco or withdrawal > 15 years
* Patient on long-term oxygen therapy
* Metal implants (thorax, spine) which can cause a deterioration in the quality of the image of the low dose scanner
* Subject included in another study protocol

Ages: 55 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects aged 55 to 74, smokers with more than 20 active pack-years or weaned for less than 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Rate of population participation in PBC screening | Baseline